CLINICAL TRIAL: NCT02185131
Title: Double-blind Pilot Trial of Mirtazapine for the Treatment of Co-occurring AD/MDD.
Acronym: PT-MAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jack Cornelius, MD, PhD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R21AA022123 (NIH); 5R21AA022123-02 (NIH)
Record Dates: First submitted 2014-06-26; First posted 2014-07-09 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-03

CONDITIONS: Major Depressive Disorder; Alcohol Use Disorder
Keywords: Major Depressive Disorder; Alcohol Use Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Alcoholism | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mirtazapine (Active Comparator): Gelatin capsules mirtazapine 15 mg, 1 capsule every a.m. Medication will be increased by one capsule, to a dose of 2 capsules barring side effects, at Week 2.
  Interventions: Drug: Mirtazapine; Drug: Placebo
- Placebo (Active Comparator): Gelatin capsules Placebo capsules, identical to mirtazapine capsules, 1 capsule every a.m. Medication will be increased by one capsule to 2 capsules at Week 2, barring any side effects.
  Interventions: Drug: Mirtazapine; Drug: Placebo

INTERVENTIONS:
Drug: Mirtazapine — Gelatin capsules mirtazapine 15 mg, 1 capsule every a.m. Medication will be increased by one capsule, to a dose of 2 capsules barring side effects, at Week 2.
  Other Names: Remeron
Drug: Placebo — Gelatin capsules Placebo capsules, identical to mirtazapine capsules, 1 capsule every a.m. Medication will be increased by one capsule to 2 capsules at Week 2, barring any side effects.

SUMMARY:
Mirtazapine is a non-SSRI (selective serotonin reuptake inhibitor) medication with a unique structure and mechanism of action. Recent study results suggest that mirtazapine may be more effective and faster acting than other antidepressants. Levels of alcohol use have been shown to be associated with levels of depressive symptoms among comorbid populations. Our own recent open label pilot study suggested robust within-group efficacy for mirtazapine for decreasing both the drinking and the depressive symptoms of persons with co-occurring alcohol dependence/major depressive disorder (AD/MDD). However, no placebo control group was employed in that study, so between-group efficacy versus placebo could not be assessed. The current grant submission proposes to conduct a first double-blind, placebo-controlled study to evaluate the efficacy of mirtazapine versus placebo for decreasing the alcohol use and depressive symptoms of persons with comorbid AD/MDD. If the results of this proposed double-blind pilot trial are promising, then the effect sizes found in this proposed study will be used to help design an adequately-powered R01 treatment trial to definitively test the efficacy of mirtazapine in this comorbid population.

DETAILED DESCRIPTION:
Alcohol dependence (AD) and Major Depressive Disorder (MDD) are among the most frequent psychiatric disorders in the general population, and the co-occurrence of those disorders represents a significant public health problem. Levels of alcohol use have been shown to be associated with levels of depressive symptoms among comorbid populations. Previous medication trials with SSRI antidepressants in this comorbid population have produced disappointing results. Mirtazapine is a non-SSRI medication with a unique structure and mechanism of action. Recent study results suggest that mirtazapine may be more effective and faster acting than other antidepressants. Our own recent open label pilot study suggested robust within-group efficacy for mirtazapine for decreasing both the drinking and the depressive symptoms of AD/MDD subjects. However, no placebo control group was employed in that study, so between-group efficacy versus placebo could not be assessed. The current grant submission proposes to conduct a first double-blind, placebo-controlled pilot study to provide a preliminary assessment of the efficacy of mirtazapine versus placebo for decreasing the alcohol use and depressive symptoms of persons with comorbid AD/MDD. If the results of this proposed double-blind pilot study are promising, then the effect sizes found in this proposed study will be used to help design an adequately-powered R01 treatment trial to definitively test the efficacy of mirtazapine versus placebo in this comorbid population.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV-TR diagnosis of current alcohol dependence, confirmed by the Mini International Neuropsychiatric Interview (MINI)
* DSM-IV-TR diagnosis of current major depressive disorder, confirmed by the Mini International Neuropsychiatric Interview (MINI)

Exclusion Criteria:

* Any person who meets criteria for alcohol-induced depression
* Any psychotic disorder bipolar disorder, mental retardation, impaired cognitive functioning, or use of any psychotropic medication in the previous month
* Current Diagnostic and Statistical Manual (DSM-IV) criteria for dependence on substances other than alcohol, cannabis, nicotine, or caffeine
* Significant neurological conditions or medical conditions
* Persistent elevation of liver function enzymes indicating active liver disease (elevated t. bilirubin or elevation to three-time normal range of liver enzymes, SGOT, SGPT, or g-GTP)
* The presence of renal function impairment defined as serum creatinine >2x upper limit of normal
* Pregnancy, inability or unwillingness to use contraceptive methods
* Use of any antidepressant medication in the prior two months, or any lifetime use of mirtazapine
* Inability to read or understand study forms and agree to informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack R Cornelius, M.D., M.P.H., Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No individual subject data will be shared.

REFERENCES:
- [Background] Cornelius JR, Douaihy AB, Clark DB, Chung T, Wood DS, Daley D. Mirtazapine in Comorbid Major Depression and Alcohol Dependence: An Open-Label Trial. J Dual Diagn. 2012 Sep 1;8(3):200-204. doi: 10.1080/15504263.2012.696527. Epub 2012 Aug 8. PMID 23230395
- [Background] Cornelius JR, Chung T, Douaihy AB, Kirisci L, Glance J, Kmiec J, FitzGerald D, Wesesky MA, Salloum I. Mirtazapine in comorbid major depression and an alcohol use disorder: A double-blind placebo-controlled pilot trial. Psychiatry Res. 2016 Aug 30;242:326-330. doi: 10.1016/j.psychres.2016.06.005. Epub 2016 Jun 15. PMID 27327217

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mirtazapine | Placebo
Started | 7 | 9
Completed | 6 | 8
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mirtazapine | Placebo | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.2 (5.9) | 37.4 (9.8) | 41.3 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Drinks Per Drinking Day
Description: Level of drinking, as indicated by the number of drinks per day as recorded on the Timeline Follow-Back calendar.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: Drinks per drinking day
Arm/Group | Mirtazapine | Placebo
Number analyzed (Participants) | 6 | 8
Drinks per drinking day | 3.5 (1.6) | 4.4 (1.5)

2. Primary Outcome: Level of Depressive Symptoms
Description: Level of depressive symptoms, as indicated by the score on the Beck Depression Inventory. The Beck Depression Inventory II scoring range is as follows: 0-13 minimal depressive symptoms, 14-19 mild depressive symptoms, 20-28 moderate depressive symptoms and 29-63 severe depressive symptoms.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Mirtazapine | Placebo
Number analyzed (Participants) | 6 | 8
Units on a scale | 27.6 (7.7) | 26.1 (11.7)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from Baseline Visit through Week 12.
Arm/Group | Mirtazapine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No